CLINICAL TRIAL: NCT01674673
Title: A Long-term Observational Study on the Efficacy of SSRIs Pharmacotherapy or Combined Treatment(SSRIs Pharmacotherapy + CBT) in Panic Disorder Patients
Brief Title: A Long-term Observational Study on the Efficacy of SSRIs or Combined Treatment(SSRIs+ CBT) in Panic Disorder Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-10-130
Record Dates: First submitted 2012-08-24; First posted 2012-08-29 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2012-08

CONDITIONS: Panic Disorder
Keywords: panic disorder; SSRIs pharmacotherapy; Cognitive Behavioral therapy
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
It is known that the treatment of panic disorder with medication and psychotherapy are both effective. Representative as a treatment for panic disorder, Selective serotonin reuptake inhibitors (SSRIs) are recommended as first-line treatment of panic disorder. In general, the initial reaction rate of panic disorder medication known to be frequently stopped early recurrence 70-80% It's too early, it is recommended that the duration of drug treatment for at least one year to be long-lasting. But whether it is appropriate for the duration of drug treatment to maintain a certain extent remains controversial, and maintain the medication for more than one year, even if the long-term effects known to be approximately 50% less than beyond being negative when remission based. Meanwhile, the typical method for the treatment of panic disorder psychology, cognitive behavioral therapy (Cognitive behavioral therapy) and looked comparable to the effect of the drug in the treatment of the known, especially in recent years when the combined treatment with medication can increase the long-term treatment of sexual reported that there's has been the subject of attention.

But prospectively compare the long-term effects of these two treatments, research, especially the research about the long-term effects of the combined treatment with the drug treatment of panic disorder is very low, and almost nil is Researchers, drug treatment and the effect of the combined treatment in patients with panic disorder over two years prospective study to compare the plans were. And verification, the researchers performed only through this study by comparing the long-term effects of the combined treatment with medication combined treatment of medication to be more effective than if the reaction to the long-term treatment of panic disorder that can affect the clinical and biological factors navigate to evaluate them. In addition, long-term observational study, panic disorder patients' subjective quality of life actually improved to some extent on the map together proven to.

DETAILED DESCRIPTION:
Panic disorder SSRI medication and long-term effects of the combined treatment on the Hamilton Rating Scale more effective treatment compared with the Scale for Anxiety (HAM-A), Clinical Psychology, I try to find the law. Drug and combination therapy of panic disorder from affecting the long-term effects on clinical (demographic and economic Factors), and to check for navigation and biological factors. - Improved quality of life to some extent due to the long-term treatment of patients with panic disorder, if you want to check

2.3 Expected Effects Panic disorder in a comparative study of the long-term effects of the combined treatment with SSRI medication until now very rare, and most of the research to target Westerners, Asians to study is almost wholly lacking. Also to investigate the nature of the clinical course of panic disorder, long-term study also little or no sleep. Elapsed for the treatment of long-term treatment of panic disorder and its impact on various clinical variables to be able to figure out if, through the analysis of the results of this study, the future could be a very useful background material, used in the development of clinical care guidelines is expected. Leading researchers in various studies for panic disorder at home and abroad, and also, therefore, the results obtained in this research is very useful in the pathogenesis and in the treatment of panic disorder is expected. The results of this study will be introduced in the Domestic Society and International Society, will finally be published in major journals of SCI related.

3 Research plan 3.1 Research information and how to

- The selection of subjects Diagnosis by the DSM-IV diagnostic criteria for major panic attacks in patients with disabilities will be conducted by a clinical psychologist or psychiatrist: Mini International Neuropsychiatric Interview Plus (MINI-plus) of structured skilled diagnostic tool.

In the case of patients who were taking medication Airlines sulfur existing at least 2 weeks (hydrochloric acid flu Jade Satin scheduled to participate in a study of the existing 4 weeks) and stop taking the drug. All other prescription non-drug (herbal medicine), forbids smoking within 24 hours before the test, caffeine drink, drinking is prohibited in the state to proceed with a test is scheduled.

Treatment conditions Randomization Randomization table belonging goes: medication alone group and the combined treatment group on either side Will be determined by the SSRIs Tx group -> Korean panic disorder treatment algorithm (Korean Medication Algorithm for Panic Disorder 2008: Initial Treatment Strategies. J. C. Yang et al., 2008) according to the treatment by applying Standardized treatment is expected to be performed. Single use only, benzodiazepine (alprazolam) and tapering zolpidem use, but only occasionally, within 3 months of treatment, so that Should, in principle, (using the PRN as alprazolam available).

* Combined Tx group SSRIs Tx group, and the same drug treatment to be carried out once a week underwent 10 sessions of CBT, and, after 3 Once a month booster session is scheduled to be performed.

  - Therapists
* Treatment conducted by a psychiatrist skilled in both groups, but CBT case of a qualified clinical psychology Scholars will participate as an adjunct therapy in the treatment session.

  * Assessment Is scheduled to visit (24 months) to assess the clinical manifestations: a total of 11 times.

Visit 1: Screening & Baseline Visit 2,3,4: every visit per month. / CBT once a week about 3 months, 10 sessions of treatment Visit 5-11: every 3 months to visit / CBT Booster session in three months, once implemented

* Visit 1 (Screening & Baseline)

  * MINI-plus diagnostic tool
  * Obtaining research consent
  * Determine whether severe medical or psychiatric diseases
  * Demographic data survey (In the future, when compared to the quality of life, according to the therapeutic, marital status, educational And income levels yuksujun compensation, and demographic and economic variables according to the comparison of the response to treatment in order) Age of onset (early onset and late-onset separated) survey
  * Clinical data (Baseline severity and panic frequency) survey

    * Duration of disease survey A comorbidity (need to MINI-plus disease confirmed) Whether other drugs: Prescription
    * Alcohol and substance combination presence Past medication or CBT, such as whether to perform
    * Hamilton Rating Scale for Anxiety (HAM-A), Hamilton Rating Scale for Depression (HAM-D), Clinical Global Impression-Severity (CGI-S), PDSS (Panic Disorder Severity Scale), Evaluate the PSR (Psychiatric status ratings)
    * As a self-assessment item MMPI-II, Anxiety Sensitivity Index-Revised (ASI-R), Albany Panic and Phobic Questionnaire (APPQ), WHOQOL-BREF, Stress Response Inventory (SRI) measurement
  * Clinical Response Remission rate Response rate and survey (No panic attack and PDSS scores <5 on standards)
  * Pharmacological Tx Drug administration and dosage, drug side effects, Compliance Survey
  * Anxiety-related biomarkers measured

    * CBC and lipid battery tests blood samples
    * Heart rate variability (HRV), Biofeedback (EMG, EDR, measuring peripheral skin temperature)
    * Cytokine (IL-1b, 2,6, TNF-alpha, IFN-r, IL-12 / IL-4, 10) measurements → blood samples
  * Genetic factor survey → blood samples

    * Serotonin related genes (5-HTTLPR & serotonin 2A receptor genetic polymorphism gene)
    * COMT, BDNF, DRD2, MAOA genetic polymorphism gene
  * Personality factor Psychiatrist skilled clinical interview of DSM-IV Axis II diagnosis enforcing
* Visit 2, 3, 4 (every 1 month, after 1, 2, and 3 Month)

  * Clinicians additional item (Clinical Global Impression-Improvement (CGI-I) rating)
  * Item self-assessment (MMPI-II)
  * Clinical Response
  * Pharmacological Tx History
  * Anxiety-related biomarkers measured (Visit 4, 3-month period)
* Visit 5-11 (every 3 months, after 6, 9 12, 15, 18, 21, 24 Month)

  * visit 2,3,4 same as the one measuring anxiety-related biomarker for 6 months, 12 months, 18 months, 24 months, and only at the point

    * Statistical analyses Methods of treatment: comparison between the two treatment groups for baseline anxiety severity, and status as a covariate Will be analyzed under analysis of covariance (ANCOVA) model using For comparison: two treatments according to the degree of improvement between the groups (remitters) the Cochran- It is planned to use the Mantel-Haenszel test. Personality or reaction and make a difference, according to the genetic factor gene to gene on gene interaction, and gene to environment interaction multiple regression or MDR (multidimensional reduction) using the statistical program is expected to be analyzed.
    * Plan for the subject's right to privacy and information protection Effect from September 30, 2011, in accordance with the Privacy Act, personal information collected purposes, the subject's right to privacy and information protection for subject identification is not possible to encrypt your name and personal number of participants in the study, and you want to collect personal items of information, the right description of the subjects for the duration of the protection of personal information and use, and is expected to obtain this consent. Information obtained from the study to the Clinical Trials Committee of the Food and Drug Administration to be used only for the purpose of analysis and clinical research information to connect to, and comply with the relevant provisions. The results of this trial will be published if the subject's identity will remain secret, and all relevant data will be managed under the supervision of the Principal Investigator.

3.2 Subjects plan Panic disorder patients 20 years of age or older to visit the Samsung Seoul Hospital, and the Department of Mental Health, a foreign patients, patients who agreed to participate in this study will be of. Plan the patient-specific total of 110 patients on each drug treatment group and combined treatment group, 55 patients recruited by the first year of study commences 2 years F / U to enforce the number of subjects. Which G * Power 3.0.10 version program (Erdfelder, E., Faul, F., & Buchner, A. (1996)), using the power 80%, significance level of 5%, effect size 0.6, and the case and control groups equal number allocation to treatment in panic disorder seems common rate, the percentage of Asian American about 20% and Samsung Seoul Hospital, Department of Mental Health, panic disorder patients for many years to visit when you consider that approximately 2,300 (initial 200 patients, at least), the appropriate is suggested by the number of subjects.

Subject selection criteria>

* Outpatients with panic disorder at the SMC
* PD patients who agree to participate in the clinical study
* PD patients who are over 20 years old

Subject exclusion criteria>

* PD patients who have either severe medical illnesses or other psychiatric illnesses
* PD patients who are pregnant, or lactating PD patients who have suicidal idea

3.3 Subjects for Risk / Benefit Risk: every 3, 6, 12, 18, and 24 months after treatment with at the time, be conducted sampling method is typically performed venous blood 60 ml (6 times). Accordingly, the subcutaneous blood or mild pain on the puncture site hematoma and bruising and discomfort of the byeolun.

In addition, the possible side effects be used to study aviation sulfur drugs, selective serotonin reuptake inhibitors, such as nausea, vomiting, dry mouth, dizziness, diarrhea, insomnia, somnolence, ejaculation delay or erectile impairment sexual interference and can be.

Suspended for the duration of existing drugs, on recurrence gonghwangjeung and cause a worsening of the subjects were taking the existing air sulfur drugs, if may be.

Interests: while participating in a clinical trial for two years, the state of mental health, and balance the autonomic nervous system, the degree and temperament / personality traits in the individual subjects to learn. Blood through the analysis of the primary results of a blood test before and after treatment may also be associated with various psychological tests, can receive free of charge.

4 Annual Research Plan (3-year study performed)

* 1st year (2012): Patient recruitment and conduct research
* 2nd year (2013): Studies performed
* 3rd year (2014): conduct research and data analysis

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with panic disorder at the SMC
* PD patients who agree to participate in the clinical study
* PD patients who are over 20 years old

Exclusion Criteria:

* PD patients who have either severe medical illnesses or other psychiatric illnesses
* PD patients who are pregnant, or lactating
* PD patients who have suicidal idea

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Panic disorder patients 20 years of age or older to visit the Samsung Seoul Hospital, and the Department of Mental Health, a foreign patients, patients who agreed to participate in this study will be of. Plan the patient-specific total of 100 patients on each drug treatment group and combined treatment group, 55 patients recruited by the first year of study commences 1 years F / U to enforce the number of subjects.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
PDSS | one year

CONTACTS AND LOCATIONS:
Overall Officials: BumHee BH Yu, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea